CLINICAL TRIAL: NCT06038253
Title: Relation Between Non- Alcoholic Fatty Liver Disease and Bone Mineral Density in Egyptian Adults
Brief Title: Relation Between NAFLD and BM DENSITY
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina maged helmy habib, Resident doctor, Assiut University
Other Study IDs: NAFLD and bone mineral density
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: NAFLD; Osteoporosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fibroscan — Fibroscan is device to detect degree of liver fibrosis in NAFLD patients Dexa scan device detect degree of osteoporosis in NAFLD patients
  Other Names: Dexa scan

SUMMARY:
In general NAFLD is a common denominal for a broad spectrum of damage to the liver, which can be due to hepatocyte injury, inflammatory processes and fibrosis. This is normally seen on liver biopsy and can range from milder forms (steatosis) to the more severe forms (non-alcoholic steatohepatitis (NASH), advanced fibrosis, cirrhosis and liver failure). In these patients, advanced fibrosis is the major predictor of morbidity and liver-related mortality, and an accurate diagnosis of NASH and NAFLD is mandatory .

NAFLD is closely associated with metabolic disorders, including central obesity, dyslipidaemia, hypertension, hyperglycaemia and persistent abnormalities of liver function tests. NAFLD was shown to be connected with diseases that are usually not dependent on obesity, such as sarcopenia and osteoporosis

Target of the study :

1. Clarify predictive value of fibroscan and u/s in diagnosis of NAFLD.
2. Estimate the metabolic effect of NAFLD on bone density
3. Estimate the correlation between obesity , NAFLD and BMD

DETAILED DESCRIPTION:
INTRODUCTION:

In general, the prevalence of NAFLD has increased over the last 20 years. The Middle East and South America have the highest NAFLD prevalence at 31% and 32% respectively with the lowest prevalence in Africa at 13.5% .

NAFLD is closely associated with metabolic disorders, including central obesity, dyslipidaemia, hypertension, hyperglycaemia and persistent abnormalities of liver function tests. NAFLD was shown to be connected with diseases that are usually not dependent on obesity, such as sarcopenia and osteoporosis In general NAFLD is a common denominal for a broad spectrum of damage to the liver, which can be due to hepatocyte injury, inflammatory processes and fibrosis. This is normally seen on liver biopsy and can range from milder forms (steatosis) to the more severe forms (non-alcoholic steatohepatitis (NASH), advanced fibrosis, cirrhosis and liver failure). In these patients, advanced fibrosis is the major predictor of morbidity and liver-related mortality, and an accurate diagnosis of NASH and NAFLD is mandatory .

Osteoporosis is a group of bone diseases with various causes, including general factors related to aging, obesity and sex steroid deficiency, as well as specific risk factors such as the use of glucocorticoids, reduced bone quality, and disruption of microarchitectural integrity. In most cases of osteoporosis, the reduction in bone tissue is mainly due to increased bone resorption. Osteoporosis is characterized by low bone mineral density (BMD), bone pain and easy fracture.Osteoporosis is a silent disease until fractures occur with increasing frequency, which can cause important problems and even death. In industrialized countries, 9%-38% of women and 1%-8% of men >50 years suffer from osteoporosis.

Therefore, osteoporosis is not only harmful to health but also increases the financial burden of the impacted countries.

Many studies have demonstrated that NAFLD is associated with low BMD and osteoporosis.

Liver is the source of many proteins and is the regulator of several pathways involving bone metabolism; one of the most well-known of all is vitamin D metabolism pathway. Considering the role of liver in bone metabolism, the association between NAFLD and bone abnormalities is not surprising especially with substantial supporting evidences in recent years .

Besides its role in the calcium and bone metabolism, vitamin D may also exert pleiotropic effects in many tissues. NAFLD patients were reported to have a marked reduction in serum 25(OH) vitamin D when compared with control Liver biopsy remains the current gold standard for diagnosis of NAFLD, despite limitations regarding sampling variability, invasive nature, and high cost. However, numerous non-invasive biomarkers, including mainly serum markers or imaging modalities, intend to detect the presence of steatosis, NASH or advanced fibrosis. To date, ultrasound is suggested as first-line screening tool for defining steatosis in a selected population, while diagnosis of NAFLD requires exclusion of other chronic liver disease etiology or other steatosis causes and exclusion of alcohol intake by history .

Fibro scan becomes an evidence based , transient elastography instrument For noninvasive evaluation of liver steatosis and fibrosis , fibroscan is becoming an increasing important modality in NAFLD practice , as it was recently used to identify patients eligible for NAFLD related clinical trials

Target of the study :

1. Clarify predictive value of fibroscan and u/s in diagnosis of NAFLD.
2. Estimate the metabolic effect of NAFLD on bone density
3. Estimate the correlation between obesity , NAFLD and BMD

STUDY DESIGN :

CROSS- SECTIONAL OBSERVATIONAL STUDY

Patients and methods :

1. Patients presented to obesity clinic for follow up
2. Patients presented to git clinic
3. Patients presented to fibroscan clinic for evaluation the degree of liver fibrosis and steatosis will be included in the study
4. Patients presented at radiology department for abd U.S and diagnosed accidentally fatty liver .

INCLUSION CRITERIA

1. Patients above the age of 18 y.o and premenopausal females
2. Patients showing any degree of fibrosis and steatosis .
3. Patients suffers from obesity and its complications
4. Patients with hyperlipidemia and diabetes mellitus .
5. NAFLD patients were diagnosed with an ultrasound examination or fibroscan or pathological examination to make a clear and definite diagnosis,
6. all the obese participants according to body mass index (BMI)
7. BMD was measured by dual energy X-ray absorptiometry.

Exclusion criteria :

1. Patients less than 18 y.o
2. Patients known alcohol abuser of ≥30 g/day in men or≥20 g/day in women.
3. Patients with chronic liver disease or hepatocellular carcinoma .
4. Subjects with suspected or proven any other liver disease other than NAFLD as (viral hepatitis, drug-induced liver injury, autoimmune liver disease, Wilson's disease or primary biliary cholangitis).
5. none of the subjects followed specific diets or therapeutic treatments that could influence BMD or liver function.
6. Patients with conditions known to affect bone metabolism, such as kidney, thyroid or parathyroid diseases, bone tumors
7. (iv) Postmenopausal females to avoid the increased risk of osteoporosis in those patients due to hormonal changes.

ELIGIBILITY:
Inclusion Criteria:

- INCLUSION CRITERIA

1. Patients above the age of 18 y.o and premenopausal females
2. Patients showing any degree of fibrosis and steatosis .
3. Patients suffers from obesity and its complications
4. Patients with hyperlipidemia and DM
5. NAFLD patients were diagnosed with an ultrasound examination or fibroscan or pathological examination to make a clear and definite diagnosis,
6. all the obese participants according to body mass index (BMI)
7. BMD was measured by dual energy X-ray absorptiometry.

Exclusion Criteria:

* 1- Patients less than 18 y.o 2- Patients known alcohol abuser of ≥30 g/day in men or≥20 g/day in women. 3- Patients with chronic liver disease or HCC. 4- Subjects with suspected or proven any other liver disease other than NAFLD as (viral hepatitis, drug-induced liver injury, autoimmune liver disease, Wilson's disease or primary biliary cholangitis).

  5- none of the subjects followed specific diets or therapeutic treatments that could influence BMD or liver function.

  6- Patients with conditions known to affect bone metabolism, such as kidney, thyroid or parathyroid diseases, bone tumors 7- (iv) Postmenopausal females to avoid the increased risk of osteoporosis in those patients due to hormonal changes.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: 1. Patients presented to obesity clinic for follow up
  2. Patients presented to git clinic at Alrajhi hospital
  3. Patients presented to fibroscan clinic for evaluation the degree of liver fibrosis and steatosis will be included in the study
  4. Patients presented at radiology department for abd U.S and diagnosed accidentally fatty liver .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Level of vit D level in serum in NAFLD patients | 1 year
  To study level of vit D in NAFLD patients and its relation to disease severity
Degree of osteoporosis in NAFLD patients | 1 year
  Using dexa scan to detect level of osteoporosis in NAFLD patients
Level of parathyroid hormone level in NAFLD PATIENTS | 1 year
  Level of parathyroid hormone level in NAFLD PATIENTS and its relation to disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abdelrahman alkhateeb, Professor, Study Director — Assiut University; Ahmed Mohammed mostafa ashmawy, Assistant professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sasso M, Audiere S, Kemgang A, Gaouar F, Corpechot C, Chazouilleres O, Fournier C, Golsztejn O, Prince S, Menu Y, Sandrin L, Miette V. Liver Steatosis Assessed by Controlled Attenuation Parameter (CAP) Measured with the XL Probe of the FibroScan: A Pilot Study Assessing Diagnostic Accuracy. Ultrasound Med Biol. 2016 Jan;42(1):92-103. doi: 10.1016/j.ultrasmedbio.2015.08.008. Epub 2015 Sep 19. PMID 26386476
- [Background] Ballestri S, Zona S, Targher G, Romagnoli D, Baldelli E, Nascimbeni F, Roverato A, Guaraldi G, Lonardo A. Nonalcoholic fatty liver disease is associated with an almost twofold increased risk of incident type 2 diabetes and metabolic syndrome. Evidence from a systematic review and meta-analysis. J Gastroenterol Hepatol. 2016 May;31(5):936-44. doi: 10.1111/jgh.13264. PMID 26667191
- [Result] Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-90. doi: 10.1038/nrgastro.2013.171. Epub 2013 Sep 17. PMID 24042449
- [Result] Eshraghian A. Bone metabolism in non-alcoholic fatty liver disease: vitamin D status and bone mineral density. Minerva Endocrinol. 2017 Jun;42(2):164-172. doi: 10.23736/S0391-1977.16.02587-6. Epub 2016 Dec 14. PMID 27973461
- [Result] Poggiogalle E, Donini LM, Lenzi A, Chiesa C, Pacifico L. Non-alcoholic fatty liver disease connections with fat-free tissues: A focus on bone and skeletal muscle. World J Gastroenterol. 2017 Mar 14;23(10):1747-1757. doi: 10.3748/wjg.v23.i10.1747. PMID 28348479